CLINICAL TRIAL: NCT01093599
Title: Phase 2 Randomized Trial on the Effectiveness of Mindfulness Training for Smokers, a Novel Intervention Designed to Help Smokers Quit Smoking
Brief Title: Trial on the Effectiveness of Mindfulness Training for Smokers
Acronym: MTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2009-0039; 1K23DA022471-01A1 (NIH)
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-01

CONDITIONS: Nicotine Dependence
Keywords: Smoking; Smoking cessation; Nicotine; Tobacco; Mindfulness; Meditation; MBSR; Mindfulness Training; Behavioral Intervention; Nicotine Patch; Quit Line; Phone counseling
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quit Line Only (Active Comparator): Control Participants will call the Wisconsin Tobacco Quit Line intervention including phone counseling, Quit Smoking Materials and 4 weeks of nicotine patches.
  Interventions: Behavioral: Quit Line Only
- Quit Line plus MTS (Active Comparator): Participants in the study group will receive the Quit Line intervention (talk to a Quit Line Counselor, receive quit smoking materials and get 4 weeks of nicotine patches) and also receive 4 weeks of training in mindfulness meditation through the mindfulness for smokers intervention.
  Interventions: Behavioral: Quit Line plus MTS

INTERVENTIONS:
Behavioral: Quit Line plus MTS — This provides the quit line intervention plus the Mindfulness for Smokers Intervention.
  Other Names: Study Group; Quit Line Plus Mindfulness Training for Smokers
  Arms: Quit Line plus MTS
Behavioral: Quit Line Only — The quit line only intervention includes phone counseling, Quit Smoking Materials and 4 weeks of nicotine patches.
  Other Names: Control Group
  Arms: Quit Line Only

SUMMARY:
The Mindfulness Training for Smokers study follows a randomized controlled design with 240 total participants. Both the study group and the control group will be enrolled in the Wisconsin Tobacco Quit Line and will receive four weeks of nicotine patches. The control group will receive the Quit Line intervention alone where as the study group will receive the Quit Line intervention plus the Mindfulness for Smokers Intervention. The Mindfulness for Smokers Intervention provides four weeks of instruction in mindfulness meditation followed by four weeks of participation in a weekly meditation group. The principal hypothesis for the study is that Mindfulness for Smokers plus the Quit Line will lead to significantly higher rates of smoking cessation at 6 months than the Quit Line alone.

DETAILED DESCRIPTION:
The MTS study is funded for through a five year K23 NIH training grant. The study follows a randomized controlled design with N = 240. Both the study group and the control group will be enrolled in the Wisconsin Tobacco Quit Line, will receive four weeks of nicotine patches, and receive phone based counseling through the Quit Line. The control group n = 120 will receive the Quit Line intervention alone where as the study group n = 120 will receive the Quit Line intervention plus the Mindfulness Training for Smokers (MTS) Intervention.

Mindfulness Training for Smokers provides 4 weeks of mindfulness meditation instruction followed by entry into a MTS meditation group. The total time for the study including recruitment, intervention and participant follow-up for N = 240 will be four years. The study will recruit subjects from the Dane county region through the University of Wisconsin School of Medicine and Public Health Center for Tobacco Research and Intervention (UW-CRTI). Recruitment will take place through the television and radio advertisements (appendix). In addition, the Wisconsin Quit Line web site will provide a link to the MTS study. With this link, quit line coaches will have a brief description of the study (see appendix) and will provide contact information for the study. Finally, the MTS web site (url: www.sittoquit.org) will provide basic introductory information available to the general public.

The principal hypothesis for the study is that MTS plus Quit Line will lead to significantly higher rates of smoking cessation at 6 months than use of the Quit Line alone. Secondary hypotheses is that study group compared to controls will show significant differences in questionnaire results that test distress, depression, anxiety, attentional control, mindfulness and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or over;
2. Participants must express "high" motivation to quit smoking
3. Participants must express willingness to attend "all" meetings for 2 months.
4. Smoke 5 or more cigarettes per day

Exclusion Criteria:

1. Self report of alcohol use of 4 drinks or more a night on 4 or more nights per week.
2. Self report of using chewing tobacco, snuff or cigars in the last week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Davis, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

REFERENCES:
- [Result] Davis JM, Goldberg SB, Anderson MC, Manley AR, Smith SS, Baker TB. Randomized trial on mindfulness training for smokers targeted to a disadvantaged population. Subst Use Misuse. 2014 Apr;49(5):571-85. doi: 10.3109/10826084.2013.770025. PMID 24611852
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- See also: Randomized trial on mindfulness training for smokers targeted to a disadvantaged population. — http://www.ncbi.nlm.nih.gov/pubmed/24611852

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quit Line Only | Quit Line Plus MTS
Started | 91 | 105
Completed | 59 | 59
Not Completed | 32 | 46
Not completed — Lost to Follow-up | 32 | 46

BASELINE CHARACTERISTICS:
Population: total enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Quit Line Only | Quit Line Plus MTS | Total
Number analyzed (Participants) | 91 | 105 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.95 (12.05) | 42.25 (14.53) | 41.65 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 53 | 98
  Male | 46 | 52 | 98
Region of Enrollment [Number; unit: participants]
  United States | 91 | 105 | 196

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: Smoking abstinence is measured by Carbon Monoxide Breath Testing in Controls vs Study Group subjects six months after the quit day.
Time Frame: 6 months post quit day
Population: intent to treat analysis
Measure: Number; unit: participants
Arm/Group | Quit Line Only | Quit Line Plus MTS
Number analyzed (Participants) | 91 | 105
participants | 13 | 24

2. Secondary Outcome: Changes in Self Reported Measures of Depression, Anxiety and Stress in Study Subjects vs Controls
Time Frame: 6 months post quit day
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Quit Line Only | Quit Line Plus MTS
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/105
Other Adverse Events (participants affected / at risk) | 0/91 | 0/105

LIMITATIONS AND CAVEATS:
A principal limitation of this study is that it is designed to compare MTS to a less intensive usual care therapy and as such lacks a time/intensity matched control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No